CLINICAL TRIAL: NCT03516630
Title: Single Centre, Single Dose, Randomised, Negative and Positive-controlled, Double-blind Trazodone vs. Negative Control (Placebo), Open-label vs. Positive Control (Moxifloxacin), 5-way Cross-over QT/QTc Study
Brief Title: Effects of Three Single Oral Doses of Trazodone on the QTc Interval Duration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry); eResearch Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 039PO16364; CRO-PK-16-314 (Other: CROSS Research S.A.)
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: Trazodone; QTc interval; Moxifloxacin
MeSH Terms: interventions — Trazodone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Subjects and the investigator administering the study products and collecting the data are blinded with respect to Trazodone and placebo treatments, and open with respect to moxifloxacin treatment. Trazodone and placebo final solutions for administration is prepared by an independent Pharmacist under open conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- TRZ 20 (Experimental): Product is administered as single dose in the morning, under fasting conditions. 10 drops for the dose of 20 mg is suspended in 120 mL of still mineral water. A wash-out interval of at least 7 days is required before the administration of the other doses foreseen in the study.
  Interventions: Drug: Trazodone 20 mg
- TRZ 60 (Experimental): Product is administered as single dose in the morning, under fasting conditions. 30 drops for the dose of 60 mg is suspended in 120 mL of still mineral water. A wash-out interval of at least 7 days is required before the administration of the other doses foreseen in the study.
  Interventions: Drug: Trazodone 60 mg
- TRZ 140 (Experimental): Product is administered as single dose in the morning, under fasting conditions. 70 drops for the dose of 140 mg is suspended in 120 mL of still mineral water. A wash-out interval of at least 7 days is required before the administration of the other doses foreseen in the study.
  Interventions: Drug: Trazodone 140 mg
- Placebo (Placebo Comparator): Product is administered as single dose in the morning, under fasting conditions. Trazodone-matching placebo corresponding to 70 drops is suspended in 120 mL of still mineral water. A wash-out interval of at least 7 days is required before the administration of the other doses foreseen in the study.
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Product is administered as single dose in the morning, under fasting conditions. One 400 mg tablet is swallowed (without chewing) with 240 mL of still mineral water. A wash-out interval of at least 7 days is required before the administration of the other doses foreseen in the study.
  Interventions: Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: Trazodone 20 mg — Oral drops
  Arms: TRZ 20
Drug: Trazodone 60 mg — Oral drops
  Arms: TRZ 60
Drug: Trazodone 140 mg — Oral drops
  Arms: TRZ 140
Drug: Placebo — Oral drops
  Arms: Placebo
Drug: Moxifloxacin 400mg — Tablet
  Other Names: Avalox
  Arms: Moxifloxacin

SUMMARY:
The present study has been designed to evaluate the effect of three doses of trazodone (20, 60 and 140 mg), in comparison to placebo, on the QT/QTc interval of healthy volunteers. Trazodone oral drops 6% formulation has been selected in order to evaluate the three doses using the same formulation, because the lowest available strength for the tablet formulations is 50 mg. According to the E14 guideline on the evaluation of QT/QTc interval prolongation and proarrhythmic potential of antiarrhytmic drugs, a negative control (placebo) and a positive control (moxifloxacin) will also be assessed.

DETAILED DESCRIPTION:
Twenty (20) healthy volunteers (about 50% males and 50% females) will be randomised.

Primary end-point:

* Evaluation of the relationship between the plasma concentration of trazodone (free base) and the change from baseline in QTc, placebo-adjusted and corrected for HR based on the Fridericia correction method (QTcF) method (∆∆QTcF).
* Trazodone can be declared to have no influence on QTc if the null hypothesis, that the upper bound of the two-sided 90% CI of the predicted mean placebo corrected change from baseline for QTcF is greater than 10 msec at the observed mean Cmax for the therapeutic dose of trazodone, can be rejected.

ELIGIBILITY:
Main Inclusion Criteria:

* Sex and Age: males/females, 20-50 years old inclusive
* Body mass index (BMI): 18.5-28 kg/m2 inclusive
* Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest (supine)
* Contraception and fertility (females only): females of child-bearing potential must be using at least one of the following reliable methods of contraception:

  1. Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
  2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
  3. A male sexual partner who agrees to use a male condom with spermicide
  4. A sterile sexual partner

Main Exclusion Criteria:

* ECG (12-leads, supine position): any of the following conditions: Heart rate <50 or >90 bpm; PR <120 or >200 msec; QRS >110 msec; QTcF males >430 msec, females >450 msec; Any qualitative/morphological abnormality except: sinus arrhythmia, isolated premature atrial complexes/premature ventricular complexes; T-wave/U-wave characteristics making determination of the end of the T-wave difficult such as biphasic T-waves, U-waves of width greater than 1/3 the width of the preceding T-wave
* Diseases: history of additional risk factors for torsade de pointes (e.g. heart failure, hypokalaemia, family history of long QT syndrome); history of significant renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
* Medications: any medications, including over the counter (OTC) medications and herbal products, and in particular medications that prolong the QT/QTc interval and potentially hepatotoxic drugs or hepatic/gastric enzyme inducers (i.e. phenobarbital, phenitoine, carbamazepine, chlorzoxazone and rifampicin) for 2 weeks before the start of the study and during the study duration. Hormonal contraceptives for females will be allowed
* Physical findings: clinically significant abnormal physical findings
* Laboratory analyses: clinically significant abnormal laboratory values
* Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study.
* Blood donation: blood donations for 3 months before this study
* Drug, alcohol, caffeine, tobacco: history of drug and/or alcohol dependence [alcohol abuse defined as >1 drink/day for females and >2 drinks/day for males, defined according to USDA Dietary Guidelines 2015-2020]; caffeine abuse (>5 cups coffee/tea/day) or tobacco abuse (more than 10 cigarettes/day)
* Drug test: positive result at the drug test at screening or day -1
* Alcohol test: positive alcohol breath test at day -1
* Grapefruit juice: grapefruit juice consumption within 2 weeks of the administration of the study treatments
* Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Relationship between trazodone plasma concentration and QTc | pre-dose (-0.25 hours) and at 0.0833, 0.1666, 0.3333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
  Evaluation of the relationship between the plasma concentration of trazodone (free base) and the change from baseline in QTc, placebo-adjusted and corrected for HR based on the Fridericia correction method (QTcF) method (∆∆QTcF).
Influence of trazodone on QTc | pre-dose (-0.25 hours) and at 0.0833, 0.1666, 0.3333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16 and 24 hours post-dose.
  Trazodone can be declared to have no influence on QTc if the null hypothesis, that the upper bound of the two-sided 90% CI of the predicted mean placebo corrected change from baseline for QTcF is greater than 10 msec at the observed mean Cmax for the therapeutic dose of trazodone, can be rejected.

CONTACTS AND LOCATIONS:
Locations (1):
- CROSS Research S.A., Phase I Unit,, Arzo, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tellone V, Rosignoli MT, Picollo R, Dragone P, Del Vecchio A, Comandini A, Radicioni M, Leuratti C, Calisti F. Effect of 3 Single Doses of Trazodone on QTc Interval in Healthy Subjects. J Clin Pharmacol. 2020 Nov;60(11):1483-1495. doi: 10.1002/jcph.1640. Epub 2020 Jun 2. PMID 32488885